CLINICAL TRIAL: NCT00066690
Title: A Phase III Trial Evaluating the Role of Ovarian Function Suppression and the Role of Exemestane as Adjuvant Therapies for Premenopausal Women With Endocrine Responsive Breast Cancer
Brief Title: Suppression of Ovarian Function With Either Tamoxifen or Exemestane Compared With Tamoxifen Alone in Treating Premenopausal Women With Hormone-Responsive Breast Cancer
Acronym: SOFT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ETOP IBCSG Partners Foundation (Network)
Collaborators: Breast International Group (Other); Cancer and Leukemia Group B (Network); National Cancer Institute (NCI) (NIH); NSABP Foundation Inc (Network); NCIC Clinical Trials Group (Network); North Central Cancer Treatment Group (Network); SWOG Cancer Research Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBCSG 24-02 / BIG 2-02; NCI-2009-01086 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000316456; BIG 2-02; 2004-000166-13; IBCSG-24-02 (Other: CTEP); U24CA075362 (NIH); NCT00917969 (obsolete NCT alias); NCT02140190 (obsolete NCT alias)
Record Dates: First submitted 2003-08-06; First posted 2003-08-07 (Estimated); Results first posted 2016-09-22 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Estrogen Receptor Positive Breast Cancer; Progesterone Receptor Positive Tumor; Recurrent Breast Carcinoma; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage IIA Breast Cancer; Stage IIB Breast Cancer; Stage IIIA Breast Cancer
Keywords: tamoxifen; ovarian function suppression + tamoxifen; ovarian function suppression + exemestane
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane; Ovariectomy; Radiotherapy; Radiation; Tamoxifen; Triptorelin Pamoate; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tamoxifen (Active Comparator): Tamoxifen 20mg orally daily for 5 years
  Interventions: Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Drug: Tamoxifen
- T+OFS (Experimental): Tamoxifen 20mg orally daily for 5 years plus ovarian function suppression (OFS; triptorelin (GnRH analogue) 3.75 mg by im injection q28 days for 5 years; or surgical oophorectomy; or ovarian irradiation)
  Interventions: Other: Laboratory Biomarker Analysis; Procedure: Oophorectomy; Other: Quality-of-Life Assessment; Radiation: Radiation Therapy; Drug: Tamoxifen; Drug: Triptorelin
- E+OFS (Experimental): Exemestane 25mg orally daily for 5 years plus ovarian function suppression (OFS; triptorelin (GnRH analogue) 3.75 mg by im injection q28 days for 5 years; or surgical oophorectomy; or ovarian irradiation)
  Interventions: Drug: Exemestane; Other: Laboratory Biomarker Analysis; Procedure: Oophorectomy; Other: Quality-of-Life Assessment; Radiation: Radiation Therapy; Drug: Triptorelin

INTERVENTIONS:
Drug: Exemestane — Exemestane 25mg orally daily for 5 years plus ovarian function suppression
  Other Names: Aromasin; FCE-24304
  Arms: E+OFS
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Oophorectomy — Undergo bilateral surgical oophorectomy
  Other Names: Female Castration; Ovariectomy
  Arms: E+OFS; T+OFS
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Radiation: Radiation Therapy — Undergo ovarian irradiation
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; Irradiation; RADIATION; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
  Arms: E+OFS; T+OFS
Drug: Tamoxifen — Tamoxifen 20mg orally daily for 5 years
  Other Names: Apo-Tamox; Clonoxifen; Dignotamoxi; Ebefen; Emblon; Estroxyn; Fentamox; Gen-Tamoxifen; Genox; ICI 46,474; ICI-46474; Jenoxifen; Kessar; Ledertam; Lesporene; Nolgen; Noltam; Nolvadex; Nolvadex-D; Nourytam; Novo-Tamoxifen; Novofen; Noxitem; Oestrifen; Oncotam; PMS-Tamoxifen; Soltamox; TAM; Tamax; Tamaxin; Tamifen; Tamizam; Tamofen; Tamoxasta; TAMOXIFEN CITRATE; Tamoxifeni Citras; Zemide
  Arms: T+OFS; Tamoxifen
Drug: Triptorelin — 3.75 mg by im injection q28 days for 5 years
  Other Names: 6-D-Tryptophan-LH-RH; 6-D-Tryptophanluteinizing Hormone-releasing Factor; AY-25650; CL-118,532; Decapeptyl; Detryptoreline; GnRH analogue; Trelstar Depot; Decapeptyl Depot
  Arms: E+OFS; T+OFS

SUMMARY:
RATIONALE: Estrogen can stimulate the growth of breast tumor cells. Ovarian function suppression combined with hormone therapy using tamoxifen or exemestane may fight breast cancer by reducing the production of estrogen. It is not yet known whether suppression of ovarian function plus either tamoxifen or exemestane is more effective than tamoxifen alone in preventing the recurrence of hormone-responsive breast cancer.

PURPOSE: This randomized phase III trial studies ovarian suppression with either tamoxifen or exemestane to see how well they work compared to tamoxifen alone in treating premenopausal women who have undergone surgery for hormone-responsive breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the disease-free survival, breast cancer-free interval, distant recurrence-free interval and overall survival of premenopausal women with endocrine-responsive breast cancer when treated with tamoxifen + ovarian function suppression (by triptorelin, oophorectomy, or ovarian irradiation) or exemestane + ovarian function suppression vs. tamoxifen alone. The primary comparison is ovarian function suppression with either tamoxifen or exemestane vs. tamoxifen alone.
* Compare the quality of life, including late side effects of early menopause, of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center, prior adjuvant/neoadjuvant chemotherapy (yes vs no), and number of positive axillary and/or internal mammary lymph nodes (0 vs 1 or more) and intended initial method of ovarian function suppression (triptorelin vs oophorectomy vs ovarian irradiation). Treatment duration is 5 years. Patients are followed every 3 months for 1 year, every 6 months for 5 years, and then annually thereafter. Quality of life is assessed at baseline, every 6 months for 2 years, and then annually for 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women (estradiol [E2] in the premenopausal range [according to institution parameters]) who meet the following criteria:

  * Patients who did not receive chemotherapy should be randomized within 12 weeks after definitive surgery; such patients should have estradiol (E2) in the premenopausal range following surgery; the only patients who do not require testing of estradiol (E2) to confirm premenopausal status are those who have been menstruating regularly during the 6 months prior to randomization and have not used any form of hormonal contraception or any other hormonal treatments during the 6 months prior to randomization
  * Patients who received prior adjuvant and/or neoadjuvant chemotherapy should be randomized after completing chemotherapy and within 8 months of the final dose of chemotherapy as soon as premenopausal status is confirmed; all such patients should have premenopausal status confirmed by an estradiol (E2) in the premenopausal range between 2 weeks and 8 months after completing chemotherapy
  * Adjuvant trastuzumab (Herceptin ®) is allowable, and is not considered to be chemotherapy for eligibility timing determination
  * Patients with temporary chemotherapy-induced amenorrhea who regain premenopausal status within eight months of the final dose of chemotherapy are eligible; (please note that some patients taking tamoxifen or aromatase inhibitors, even without evidence of menses, may have ovarian function recovery following chemotherapy and resume estradiol secretion); in patients wishing to participate in the study, with postmenopausal hormone levels shortly after chemotherapy, it is recommended to recheck their estradiol level at a later timepoint within 8 months of completing chemotherapy, even in the absence of return of menses
* Histologically proven, resected breast cancer; pathology material should be available for submission for central review as part of the quality control measures for this protocol
* Patients must have hormone receptor positive tumors; if there is more than one breast tumor, each tumor must be hormone receptor positive; hormone receptors must be determined using immunohistochemistry; estrogen receptor (ER) and/or progesterone receptor (PgR) must be greater than or equal to 10% of the tumor cells positive by immunohistochemical evaluation; biochemical determination alone is not acceptable
* The tumor must be confined to the breast and axillary nodes without detected metastases elsewhere, with the exception of tumor detected in internal mammary chain nodes by sentinel node procedure; patients who received neoadjuvant therapy must have had operable disease prior to neoadjuvant treatment to be eligible; patients who had a pathological evaluation with tru cut or core biopsy of invasive breast cancer prior to neoadjuvant therapy and were found to have no invasive tumor in the pathological specimen from definitive surgery are eligible; for these patients, pre-neoadjuvant tumor characteristics will be used for defining eligibility; in case of persistent disease, pathology findings from the definitive surgery should be used
* Patients must have had proper surgery for primary breast cancer with no known clinical residual loco-regional disease:

  * A total mastectomy; radiotherapy is optional after mastectomy OR
  * A breast-conserving procedure (lumpectomy, quadrantectomy or partial mastectomy with margins clear of invasive cancer and ductal breast carcinoma in situ [DCIS]); the local pathologist must document negative margins of resection in the pathology report; if all other margins are clear, a positive posterior (deep) margin is permitted, provided the surgeon documents that the excision was performed down to the pectoral fascia and all tumor has been removed; likewise, if all other margins are clear, a positive anterior (superficial; abutting skin) margin is permitted provided the surgeon documents that all tumor has been removed; radiation therapy to the conserved breast is required; patients may be randomized before, during or after completion of radiation therapy to the breast
* Either axillary lymph node dissection (pathological examination of at least 6 nodes recommended) or a negative axillary sentinel node biopsy (pN0[sn]) is required; patients with negative or microscopically axillary positive sentinel nodes (pN1mi: micrometastasis none > 2.0 mm) do not require further axillary therapy; those with positive sentinel nodes must have either an axillary dissection or radiation of axillary nodes
* For International Breast Cancer Study Groups (IBCSG) centers, patients must have completed baseline Quality of Life (QL) Forms prior to randomization; the only exceptions are cognitive or physical impairment that interferes with QL assessment or inability to read any of the languages available on IBCSG QL forms; for non-IBCSG centers, extent of participation in the QL study is to be determined at the activation of the trial for each cooperative group
* Written informed consent must be signed and dated by the patient and the investigator prior to randomization
* Patients must be accessible for follow-up
* Patients must be informed of and agree to data and tissue material transfer and handling, in accordance with national data protection guidelines

Exclusion Criteria:

* Patients who are postmenopausal (i.e., do not have an estradiol [E2] level in the premenopausal range) after surgery or after chemotherapy, whichever is later
* Patients with distant metastatic disease
* Patients with locally advanced inoperable breast cancer including inflammatory breast cancer or supraclavicular node involvement or with enlarged internal mammary nodes (unless pathologically negative) are not eligible; patients with involved internal mammary nodes detected by sentinel node biopsy that are not enlarged are eligible
* Patients with positive final margins (referring to only DCIS and invasive cancer, not lobular breast carcinoma in situ [LCIS]), except as noted; DCIS at a margin is permitted if a complete mastectomy has been performed
* Patients with clinically detectable residual axillary disease
* Patients with a history of prior ipsilateral or contralateral invasive breast cancer; patients with synchronous bilateral invasive breast cancer (diagnosed histologically within 2 months) are eligible if the bilateral disease meets all other eligibility criteria
* Patients with previous or concomitant invasive malignancy are not eligible; the exceptions are patients with the following (and only the following) malignancies (previous or concomitant) who are eligible if adequately treated:

  * Basal or squamous cell carcinoma of the skin
  * In situ non-breast carcinoma without invasion
  * Contra- or ipsilateral in situ breast carcinoma
  * Non-breast invasive malignancy diagnosed at least 5 years ago and without recurrence:

    * Stage I papillary thyroid cancer
    * Stage Ia carcinoma of the cervix
    * Stage Ia or b endometrioid endometrial cancer
    * Borderline or stage I ovarian cancer
* Patients with other non-malignant systemic diseases (cardiovascular, renal, hepatic, lung, etc.) that would prevent prolonged follow-up; patients with previous thrombosis (e.g., deep vein thrombosis [DVT]) and/or embolism can be included only if medically suitable
* Patients who have had a bilateral oophorectomy or ovarian irradiation; patients who will be recommended to undergo oophorectomy within 5 years (e.g., breast cancer susceptibility gene [BRCA]1/2 gene carriers) and therefore for whom randomization to a treatment arm without OFS is inappropriate
* Patients with a history of noncompliance to medical regimens and patients who are considered potentially unreliable
* Patients who are pregnant or lactating at the time of randomization or who desire a pregnancy within 5 years; patients planning to use additional hormonal therapy apart from the randomized treatment during the next five years including all types of hormonal contraception; a pregnancy test is recommended for women of child-bearing potential who are sexually active and not using reliable contraceptive methods
* Patients who received endocrine therapy (including neoadjuvant and adjuvant) for more than 8 months after their breast cancer diagnosis; patients who are receiving endocrine therapy at randomization (and have received it for less than 8 months) may continue such therapy until protocol-specified tamoxifen/exemestane is initiated
* Patients who were taking tamoxifen or other selective estrogen receptor modulator (SERM) (e.g. Raloxifene) or hormone replacement therapy (HRT) within one year prior to their breast cancer diagnosis; prior oral contraceptives are allowed
* Patients who have received GnRH analogues as part of their breast cancer treatment prior to randomization
* Patients with psychiatric, addictive, or any disorder that would prevent compliance with protocol requirements

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3066 (Actual)
Dates: Start 2003-12-17 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2024-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gini Fleming, Principal Investigator — ETOP IBCSG Partners Foundation
Locations (500):
- United States (480):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Mills - Peninsula Hospitals, Burlingame, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Valley Medical Oncology Consultants-Castro Valley, Castro Valley, California
  - John Muir Medical Center-Concord Campus, Concord, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Valley Medical Oncology Consultants-Fremont, Fremont, California
  - Glendale Memorial Hospital and Health Center, Glendale, California
  - Marin General Hospital, Greenbrae, California
  - Scripps Cancer Center, La Jolla, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Memorial Medical Center, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Bay Area Tumor Institute, Oakland, California
  - Hematology and Oncology Associates-Oakland, Oakland, California
  - Tom K Lee Inc, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute, Palo Alto, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Mercy Regional Cancer Center, Redding, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Mercy General Hospital, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - Salinas Valley Memorial, Salinas, California
  - University of California San Diego, San Diego, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Veterans Administration-San Diego Medical Center, San Diego, California
  - San Francisco General Hospital, San Francisco, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Santa Rosa Memorial Hospital, Sana Rosa, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Memorial Hospital Colorado Springs, Colorado Springs, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Denver Veterans Administration Medical Center, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program NCORP, Denver, Colorado
  - The Shaw Regional Cancer Center, Edwards, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Stamford Hospital/Bennett Cancer Center, Stamford, Connecticut
  - Charlotte Hungerford Hospital Center for Cancer Care, Torrington, Connecticut
  - Bayhealth Medical Center at Kent General, Dover, Delaware
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Nanticoke Memorial Hospital, Seaford, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Cancer Research Network Inc, Boca Raton, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Cancer Specialists - Sarasota Downtown, Sarasota, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Atlanta Regional CCOP, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - Augusta Oncology Associates PC-Saint Sebastian, Augusta, Georgia
  - Well Star Cobb Hospital, Austell, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Dekalb Medical Center, Decatur, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Harbin Clinic Medical Oncology and Clinical Research, Rome, Georgia
  - Memorial University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex - Hospital, Hopedale, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - OSF Saint Anthony Medical Center, Rockford, Illinois
  - Sarah Culbertson Memorial Hospital, Rushville, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Community Hospital East, Indianapolis, Indiana
  - Community Regional Cancer Care-North, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - IU Health Arnett Cancer Care, Lafayette, Indiana
  - Horizon Oncology Center, Lafayette, Indiana
  - Saint Joseph Regional Medical Center - Mishawaka, Mishawaka, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Saint Luke's Hospital, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Genesis Medical Center - East Campus, Davenport, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Finley Hospital, Dubuque, Iowa
  - Medical Associates Clinic PC, Dubuque, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Memorial Hospital of Arkansas City, Arkansas City, Kansas
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Saint Francis Hospital and Medical Center - Topeka, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Main Office, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Louisiana State University Health Sciences Center Shreveport, Shreveport, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Mercy Hospital, Portland, Maine
  - Anne Arundel Medical Center, Annapolis, Maryland
  - Harbor Hospital Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Suburban Hospital, Bethesda, Maryland
  - Union Hospital of Cecil County, Elkton MD, Maryland
  - Kaiser Permanente - Largo Medical Center, Largo, Maryland
  - Kaiser Permanente - Towson Medical Center, Lutherville, Maryland
  - Kaiser Permanente - Shady Grove Medical Center, Rockville, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Brigham and Women's Faulkner Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Emerson Hospital/MGH Cancer Center, Concord, Massachusetts
  - Mass General/North Shore Cancer Center, Danvers, Massachusetts
  - MetroWest Medical Center-Framingham Union Hospital, Framingham, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - South Shore Hospital, South Weymouth, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Marquette General Hospital, Marquette, Michigan
  - Mid-Michigan Medical Center - Midland, Midland, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Saint Joseph's Hospital - Healtheast, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology and Hematology PA-Woodbury, Woodbury, Minnesota
  - Woodwinds Health Campus, Woodbury, Minnesota
  - Keesler Medical Center, Kessler Air Force Base, Mississippi
  - Mercy Hospital Springfield, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Saint Anthony's Medical Center, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Benefis Healthcare-West Campus, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Renown Regional Medical Center, Reno, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Exeter Hospital, Exeter, New Hampshire
  - New Hampshire Oncology Hematology PA-Hooksett, Hooksett, New Hampshire
  - Cheshire Medical Center-Dartmouth-Hitchcock Keene, Keene, New Hampshire
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Elliot Hospital, Manchester, New Hampshire
  - Frisbie Hospital, Rochester, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - The Cancer Institute of New Jersey Hamilton, Hamilton, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Hematology Oncology Associates, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Kings County Hospital, Brooklyn, New York
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - University Hospital of Brooklyn, Brooklyn, New York
  - Brookdale Hospital Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Adirondack Cancer Center, Glens Falls, New York
  - Northwell Health NCORP, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Saint Vincent's Hospital and Medical Center of New York, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Staten Island University Hospital, Staten Island, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Mission Hospital-Memorial Campus, Asheville, North Carolina
  - Hope Women's Cancer Centers-Asheville, Asheville, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas HealthCare System NorthEast, Concord, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hosiptal, Pinehurst, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Southeast Clinical Oncology Research (SCOR) Consortium NCORP, Winston-Salem, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Altru Hospital, Grand Forks, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Flower Hospital, Sylvania, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Tod Children's Hospital - Forum Health, Youngstown, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Bend Memorial Clinic, Bend, Oregon
  - Saint Charles Medical Center-Bend, Bend, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Western Oncology Research Consortium, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Hershey Cancer Institute-Clinical Trials Office, Hershey, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Saint Mary Medical and Regional Cancer Center, Langhorne, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Aria Health-Torresdale Campus, Philadelphia, Pennsylvania
  - Chestnut Hill Health System, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Scranton Hematology Oncology, Scranton, Pennsylvania
  - Grand View Hospital, Sellersville, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Women and Infants Hospital, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island
  - AnMed Health Hospital, Anderson, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Sanford Cancer Center-Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Memorial Hospital, Chattanooga, Tennessee
  - Jones Clinic, Germantown, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Nashville Oncology Associates PC, Nashville, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Medical City Dallas Hospital, Dallas, Texas
  - Zale Lipshy University Hospital, Dallas, Texas
  - Clements University Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Doctor's Hospital of Laredo, Laredo, Texas
  - Covenant Medical Center-Lakeside, Lubbock, Texas
  - Cancer Therapy and Research Center at The UT Health Science Center at San Antonio, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Southwestern Vermont Medical Center, Bennington, Vermont
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont College of Medicine, Burlington, Vermont
  - Kaiser Permanente - Fair Oaks Medical Center, Fairfax, Virginia
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - MultiCare Auburn Medical Center, Auburn, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Providence - Saint Peter Hospital, Olympia, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Group Health Cooperative of Puget Sound Oncology Consortium, Seattle, Washington
  - Group Health Cooperative-Seattle, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - MultiCare Allenmore Hospital, Tacoma, Washington
  - Northwest NCI Community Oncology Research Program, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - Multicare Health System, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Sacred Heart Hospital, Eau Claire, Wisconsin
  - Midelfort Clinic-Clairemont Campus, Eau Claire, Wisconsin
  - Aurora Cancer Care-Southern Lakes, Elkhorn, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Mary's Hospital, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - UW Health Oncology-One South Park, Madison, Wisconsin
  - Dean Hematology and Oncology Clinic, Madison, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Vince Lombardi Cancer Clinic-Marinette, Marinette, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Medical Consultants Limited, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
- Canada (19):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA-Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - Penticton Regional Hospital, Penticton, British Columbia
  - BCCA-Fraser Valley Cancer Centre, Surrey, British Columbia
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Doctor H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - Health Sciences North, Greater Sudbury, Ontario
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - London Regional Cancer Program, London, Ontario
  - Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario
  - Thunder Bay Regional Health Science Centre, Thunder Bay, Ontario
  - Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario
  - CSSS Champlain-Charles Le Moyne, Greenfield Park, Quebec
  - CHUM-Hotel Dieu du Montreal, Montreal, Quebec
  - Hopital Du Sacre-Coeur de Montreal, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
- International Breast Cancer Study Group, Bern, Switzerland

REFERENCES:
- [Result] Francis PA, Regan MM, Fleming GF, Lang I, Ciruelos E, Bellet M, Bonnefoi HR, Climent MA, Da Prada GA, Burstein HJ, Martino S, Davidson NE, Geyer CE Jr, Walley BA, Coleman R, Kerbrat P, Buchholz S, Ingle JN, Winer EP, Rabaglio-Poretti M, Maibach R, Ruepp B, Giobbie-Hurder A, Price KN, Colleoni M, Viale G, Coates AS, Goldhirsch A, Gelber RD; SOFT Investigators; International Breast Cancer Study Group. Adjuvant ovarian suppression in premenopausal breast cancer. N Engl J Med. 2015 Jan 29;372(5):436-46. doi: 10.1056/NEJMoa1412379. Epub 2014 Dec 11. PMID 25495490
- [Result] Francis PA, Fleming GF, Lang I, Ciruelos EM, Bonnefoi HR, Bellet M, Bernardo A, Climent MA, Martino S, Bermejo B, Burstein HJ, Davidson NE, Geyer CE Jr, Walley BA, Ingle JN, Coleman RE, Muller B, Le Du F, Loibl S, Winer EP, Ruepp B, Loi S, Colleoni M, Coates AS, Gelber RD, Goldhirsch A, Regan MM; SOFT Investigators and the International Breast Cancer Study Group (a division of ETOP IBCSG Partners Foundation). Adjuvant Endocrine Therapy in Premenopausal Breast Cancer: 12-Year Results From SOFT. J Clin Oncol. 2023 Mar 1;41(7):1370-1375. doi: 10.1200/JCO.22.01065. Epub 2022 Dec 9. PMID 36493334
- [Derived] O'Regan RM, Ren Y, Zhang Y, Fleming GF, Francis PA, Pagani O, Walley BA, Kammler R, Dell'Orto P, Viale G, Loi S, Colleoni M, Treuner K, Regan MM. Identifying premenopausal patients with early-stage hormone receptor-positive breast cancer at minimal risk of distant recurrence by breast cancer index. Breast. 2026 Jan 29;86:104714. doi: 10.1016/j.breast.2026.104714. Online ahead of print. PMID 41637791
- [Derived] Ribi K, Cole BF, Fleming GF, Walley BA, Francis PA, Abdi E, Burstein HJ, Cheng KL, Chia SKL, Dakhil SR, Davidson NE, Della-Fiorentina SA, Frith AE, Levine E, Lupichuk S, Pritchard K, Salim M, Stearns V, Stewart J, Valero V, van der Westhuizen A, Pagani O, Loi S, Colleoni M, Gelber RD, Goldhirsch A, Coates AS, Regan MM, Bernhard J. Prognostic value of patient-reported depression in women with hormone-responsive early breast cancer in TEXT and SOFT. Cancer. 2025 Oct 1;131(19):e70094. doi: 10.1002/cncr.70094. PMID 40986647
- [Derived] Pagani O, Walley BA, Fleming GF, Colleoni M, Lang I, Gomez HL, Tondini C, Burstein HJ, Goetz MP, Ciruelos EM, Stearns V, Bonnefoi HR, Martino S, Geyer CE Jr, Chini C, Puglisi F, Spazzapan S, Ruhstaller T, Winer EP, Ruepp B, Loi S, Coates AS, Gelber RD, Goldhirsch A, Regan MM, Francis PA; SOFT and TEXT Investigators and the International Breast Cancer Study Group (a division of ETOP IBCSG Partners Foundation). Adjuvant Exemestane With Ovarian Suppression in Premenopausal Breast Cancer: Long-Term Follow-Up of the Combined TEXT and SOFT Trials. J Clin Oncol. 2023 Mar 1;41(7):1376-1382. doi: 10.1200/JCO.22.01064. Epub 2022 Dec 15. PMID 36521078
- [Derived] Pagani O, Francis PA, Fleming GF, Walley BA, Viale G, Colleoni M, Lang I, Gomez HL, Tondini C, Pinotti G, Di Leo A, Coates AS, Goldhirsch A, Gelber RD, Regan MM; SOFT and TEXT Investigators and International Breast Cancer Study Group. Absolute Improvements in Freedom From Distant Recurrence to Tailor Adjuvant Endocrine Therapies for Premenopausal Women: Results From TEXT and SOFT. J Clin Oncol. 2020 Apr 20;38(12):1293-1303. doi: 10.1200/JCO.18.01967. Epub 2019 Oct 16. PMID 31618131
- [Derived] Francis PA, Pagani O, Fleming GF, Walley BA, Colleoni M, Lang I, Gomez HL, Tondini C, Ciruelos E, Burstein HJ, Bonnefoi HR, Bellet M, Martino S, Geyer CE Jr, Goetz MP, Stearns V, Pinotti G, Puglisi F, Spazzapan S, Climent MA, Pavesi L, Ruhstaller T, Davidson NE, Coleman R, Debled M, Buchholz S, Ingle JN, Winer EP, Maibach R, Rabaglio-Poretti M, Ruepp B, Di Leo A, Coates AS, Gelber RD, Goldhirsch A, Regan MM; SOFT and TEXT Investigators and the International Breast Cancer Study Group. Tailoring Adjuvant Endocrine Therapy for Premenopausal Breast Cancer. N Engl J Med. 2018 Jul 12;379(2):122-137. doi: 10.1056/NEJMoa1803164. Epub 2018 Jun 4. PMID 29863451
- [Derived] Regan MM, Walley BA, Francis PA, Fleming GF, Lang I, Gomez HL, Colleoni M, Tondini C, Pinotti G, Salim M, Spazzapan S, Parmar V, Ruhstaller T, Abdi EA, Gelber RD, Coates AS, Goldhirsch A, Pagani O. Concurrent and sequential initiation of ovarian function suppression with chemotherapy in premenopausal women with endocrine-responsive early breast cancer: an exploratory analysis of TEXT and SOFT. Ann Oncol. 2017 Sep 1;28(9):2225-2232. doi: 10.1093/annonc/mdx285. PMID 28911092
- [Derived] Regan MM, Francis PA, Pagani O, Fleming GF, Walley BA, Viale G, Colleoni M, Lang I, Gomez HL, Tondini C, Pinotti G, Price KN, Coates AS, Goldhirsch A, Gelber RD. Absolute Benefit of Adjuvant Endocrine Therapies for Premenopausal Women With Hormone Receptor-Positive, Human Epidermal Growth Factor Receptor 2-Negative Early Breast Cancer: TEXT and SOFT Trials. J Clin Oncol. 2016 Jul 1;34(19):2221-31. doi: 10.1200/JCO.2015.64.3171. Epub 2016 Apr 4. PMID 27044936
- [Derived] Ribi K, Luo W, Bernhard J, Francis PA, Burstein HJ, Ciruelos E, Bellet M, Pavesi L, Lluch A, Visini M, Parmar V, Tondini C, Kerbrat P, Perello A, Neven P, Torres R, Lombardi D, Puglisi F, Karlsson P, Ruhstaller T, Colleoni M, Coates AS, Goldhirsch A, Price KN, Gelber RD, Regan MM, Fleming GF. Adjuvant Tamoxifen Plus Ovarian Function Suppression Versus Tamoxifen Alone in Premenopausal Women With Early Breast Cancer: Patient-Reported Outcomes in the Suppression of Ovarian Function Trial. J Clin Oncol. 2016 May 10;34(14):1601-10. doi: 10.1200/JCO.2015.64.8675. Epub 2016 Mar 28. PMID 27022111
- [Derived] Bernhard J, Luo W, Ribi K, Colleoni M, Burstein HJ, Tondini C, Pinotti G, Spazzapan S, Ruhstaller T, Puglisi F, Pavesi L, Parmar V, Regan MM, Pagani O, Fleming GF, Francis PA, Price KN, Coates AS, Gelber RD, Goldhirsch A, Walley BA. Patient-reported outcomes with adjuvant exemestane versus tamoxifen in premenopausal women with early breast cancer undergoing ovarian suppression (TEXT and SOFT): a combined analysis of two phase 3 randomised trials. Lancet Oncol. 2015 Jul;16(7):848-58. doi: 10.1016/S1470-2045(15)00049-2. Epub 2015 Jun 16. PMID 26092816
- [Derived] Pagani O, Regan MM, Walley BA, Fleming GF, Colleoni M, Lang I, Gomez HL, Tondini C, Burstein HJ, Perez EA, Ciruelos E, Stearns V, Bonnefoi HR, Martino S, Geyer CE Jr, Pinotti G, Puglisi F, Crivellari D, Ruhstaller T, Winer EP, Rabaglio-Poretti M, Maibach R, Ruepp B, Giobbie-Hurder A, Price KN, Bernhard J, Luo W, Ribi K, Viale G, Coates AS, Gelber RD, Goldhirsch A, Francis PA; TEXT and SOFT Investigators; International Breast Cancer Study Group. Adjuvant exemestane with ovarian suppression in premenopausal breast cancer. N Engl J Med. 2014 Jul 10;371(2):107-18. doi: 10.1056/NEJMoa1404037. Epub 2014 Jun 1. PMID 24881463
- [Derived] Regan MM, Pagani O, Fleming GF, Walley BA, Price KN, Rabaglio M, Maibach R, Ruepp B, Coates AS, Goldhirsch A, Colleoni M, Gelber RD, Francis PA; International Breast Cancer Study; GroupSOFT and TEXT Investigators. Adjuvant treatment of premenopausal women with endocrine-responsive early breast cancer: design of the TEXT and SOFT trials. Breast. 2013 Dec;22(6):1094-100. doi: 10.1016/j.breast.2013.08.009. Epub 2013 Oct 2. PMID 24095609

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 3066 patients were randomized between 17Dec03 and 27Jan11 at 426 centers in 25 countries.
Period: Overall Study
Arm/Group | Tamoxifen | T+OFS | E+OFS
Started | 1021 | 1024 | 1021
Completed | 654 | 751 | 719
Not Completed | 367 | 273 | 302
Not completed — Adverse Event | 146 | 70 | 135
Not completed — Death | 3 | 0 | 2
Not completed — Lack of Efficacy | 114 | 113 | 77
Not completed — Lost to Follow-up | 50 | 33 | 39
Not completed — Withdrawal by Subject | 54 | 57 | 49

BASELINE CHARACTERISTICS:
Population: Intention-to-treat population, excludes 19 patients who immediately withdrew consent.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tamoxifen | T+OFS | E+OFS | Total
Number analyzed (Participants) | 1018 | 1015 | 1014 | 3047
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 43 [38 to 46] | 43 [38 to 47] | 43 [38 to 47] | 43 [38 to 47]
Sex/Gender, Customized [Number; unit: percent of participants] — Units in this baseline measure reflect the percentage of total participants, rather than number of participants. The total provided does not equal the total number of participants and should not be interpreted as an accurate total of participants.
  percent of participants
    Female | 100 | 100 | 100 | 300
    Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaskan native | 1 | 5 | 3 | 9
  Asian | 36 | 34 | 33 | 103
  Black/African American | 32 | 27 | 34 | 93
  Hawaiian/Pacific Islander | 5 | 4 | 3 | 12
  White/Caucasian | 877 | 873 | 866 | 2616
  Other | 4 | 2 | 3 | 9
  Unknown | 19 | 22 | 22 | 63
  Hispanic/Latino/South American native | 44 | 48 | 50 | 142
Lymph-node status [Number; unit: percent of participants] — Units in this baseline measure reflect the percentage of total participants, rather than number of participants. The total provided does not equal the total number of participants and should not be interpreted as an accurate total of participants.
  percent of participants
    Negative | 65.03 | 65.22 | 66.17 | 196.42
    Positive | 34.97 | 34.78 | 33.83 | 103.58
Tumor size [Number; unit: percent of participants] — Units in this baseline measure reflect the percentage of total participants, rather than number of participants. The total provided does not equal the total number of participants and should not be interpreted as an accurate total of participants.
  percent of participants
    Unknown | 2.65 | 2.46 | 2.07 | 7.18
    <=2 cm | 66.40 | 64.63 | 66.86 | 197.89
    >2cm | 30.94 | 32.91 | 31.07 | 94.92
Tumor grade [Number; unit: percent of participants] — Tumor grade is the histologic grade according to the BRE method. The method involves assessment of tumor morphology, including tubule formation, nuclear pleomorphism and frequency of mitoses. Grades are recorded according to criteria as 1,2 or 3. Grade 3 is associated with poor prognosis.
  Units in this baseline measure reflect the percentage of total participants, rather than number of participants. The total provided does not equal the total number of participants and should not be interpreted as an accurate total of participants.
  percent of participants
    Unknown | 2.36 | 2.36 | 2.17 | 6.89
    1 | 27.01 | 26.11 | 24.36 | 77.48
    2 | 48.33 | 50.64 | 53.65 | 152.62
    3 | 22.30 | 20.89 | 19.82 | 63.01
HER2-status [Number; unit: percent of participants] — Units in this baseline measure reflect the percentage of total participants, rather than number of participants. The total provided does not equal the total number of participants and should not be interpreted as an accurate total of participants.
  percent of participants
    Unknown | 4.32 | 2.86 | 2.66 | 9.84
    Negative | 84.18 | 85.42 | 84.52 | 254.12
    Positive | 11.49 | 11.72 | 12.82 | 36.03

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival
Description: Estimated percentage of patients alive and disease-free at 5 years from randomization, where disease-free survival is defined as the time from randomization to the first appearance of one of the following: invasive breast cancer recurrence at local, regional, or distant site, invasive contralateral breast cancer, second (non-breast) invasive cancer, or death without cancer event; or censored at date of last follow-up.
Time Frame: 5-year estimates, reported at a median follow-up of 67 months.
Population: Intention-to-treat
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tamoxifen | T+OFS | E+OFS
Number analyzed (Participants) | 1018 | 1015 | 1014
percentage of participants | 84.7 [82.2 to 86.9] | 86.6 [84.2 to 88.7] | 89 [86.8 to 90.9]
Statistical Analysis 1: Comparison: Tamoxifen vs T+OFS; Test type: Superiority; p = 0.1, Log Rank; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.66 to 1.04] — Tamoxifen was the reference group in the estimation of the hazard ratio
Statistical Analysis 2: Comparison: Tamoxifen vs E+OFS; Test type: Superiority; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.53 to 0.86] — Tamoxifen was the reference group in the estimation of the hazard ratio

2. Secondary Outcome: Breast Cancer-free Interval
Description: Estimated percentage of patients alive and disease-free at 5 years from randomization, where breast cancer-free interval is defined as the time from randomization to invasive breast cancer recurrence at local, regional, or distant site, or invasive contralateral breast cancer; or censored at date of last follow up.
Time Frame: 5-year estimates, reported at a median follow-up of 67 months.
Population: Intention-to-treat
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tamoxifen | T+OFS | E+OFS
Number analyzed (Participants) | 1018 | 1015 | 1014
percentage of participants | 86.4 [84.0 to 88.5] | 88.4 [86.1 to 90.3] | 90.9 [88.9 to 92.6]
Statistical Analysis 1: Comparison: Tamoxifen vs T+OFS; Test type: Superiority; p = 0.09, Log Rank; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.3 to 1.03] — Tamoxifen was the reference group in the estimation of the hazard ratio
Statistical Analysis 2: Comparison: Tamoxifen vs E+OFS; Test type: Superiority; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.49 to 0.83] — Tamoxifen was the reference group in the estimation of the hazard ratio

3. Secondary Outcome: Distant Recurrence-free Interval
Description: Estimated percentage of patients alive and disease-free at 5 years from randomization, where distant recurrence-free Interval is defined as the time from randomization to invasive breast cancer recurrence at distant site, or invasive contralateral breast cancer; or censored at date of last follow up.
Time Frame: 5-year estimates, reported at a median follow-up of 67 months.
Population: Intention-to-treat
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tamoxifen | T+OFS | E+OFS
Number analyzed (Participants) | 1018 | 1015 | 1014
percentage of participants | 90.7 [88.6 to 92.4] | 91.3 [89.2 to 92.9] | 93.0 [91.2 to 94.5]
Statistical Analysis 1: Comparison: Tamoxifen vs T+OFS; Test type: Superiority; p = 0.40, Log Rank; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.66 to 1.18] — T was the reference group in the estimation of the hazard ratio
Statistical Analysis 2: Comparison: Tamoxifen vs E+OFS; Test type: Superiority; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.52 to 0.96] — T was the reference group in the estimation of hazard ratio

4. Secondary Outcome: Overall Survival
Description: Estimated percentage of patients alive at 8 years from randomization, where overall survival is defined as the time from randomization to death from any cause; or censored at date last known alive.
Time Frame: 8-year estimates, reported at a median follow-up of 8 years
Population: Intention-to-treat
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tamoxifen | T+OFS | E+OFS
Number analyzed (Participants) | 1018 | 1015 | 1014
percentage of participants | 91.5 [89.4 to 93.2] | 93.3 [91.4 to 94.8] | 92.1 [90.0 to 93.7]
Statistical Analysis 1: Comparison: Tamoxifen vs T+OFS; Test type: Superiority — [not specified]; p = 0.01, Log Rank; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.48 to 0.92] — T was the reference group in the estimation of the hazard ratio
Statistical Analysis 2: Comparison: Tamoxifen vs E+OFS; Test type: Superiority — [not specified]; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.62 to 1.15] — T was the reference group in the estimation of hazard ratio

ADVERSE EVENTS:
Time Frame: Assessed every 3 months for the first year, then every 6 month until year 6. Reported at a median follow-up of 67 months.
Description: Targeted AEs and other grade 3 or higher AEs were collected on CRFs, regardless of attribution. The safety population EXCLUDES patients who never started protocol-assigned therapy.
Arm/Group | Tamoxifen | T+OFS | E+OFS
All-Cause Mortality (participants affected / at risk) | 87/1007 | 68/1007 | 80/1001
Serious Adverse Events (participants affected / at risk) | 315/1007 | 375/1007 | 375/1001
Other Adverse Events (participants affected / at risk) | 951/1007 | 982/1007 | 980/1001
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tamoxifen (N=1007) | T+OFS (N=1007) | E+OFS (N=1001)
Hemoglobin (Blood and lymphatic system disorders) | 2 | 2 | 2
Cardiac Arrhythmia-Other (Specify) (Cardiac disorders) | 0 | 1 | 0
Cardiac-ischemia/infarction (Cardiac disorders) | 4 | 1 | 3
Conduction abnormality/Atrioventricular heart block - AV block-third degree (complete AV block) (Cardiac disorders) | 0 | 0 | 1
Conduction abnormality/Atrioventricular heart block - Sick sinus syndrome (Cardiac disorders) | 0 | 0 | 1
Left ventricular diastolic dysfunction (Cardiac disorders) | 0 | 0 | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 2 | 3
Pain - Cardiac/heart (Cardiac disorders) | 0 | 0 | 1
Restrictive cardiomyopathy (Cardiac disorders) | 0 | 0 | 1
Right ventricular dysfunction (cor pulmonale) (Cardiac disorders) | 0 | 0 | 1
Supraventricular and nodal arrhythmia - Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Supraventricular and nodal arrhythmia - Sinus arrhythmia (Cardiac disorders) | 0 | 1 | 0
Supraventricular and nodal arrhythmia - Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Valvular heart disease (Cardiac disorders) | 2 | 0 | 0
Auditory/Ear-Other (Specify) (Ear and labyrinth disorders) | 1 | 0 | 0
Hearing: patients without baseline audiogram and not enrolled in a monitoring program (Ear and labyrinth disorders) | 1 | 0 | 1
Thyroid function, high (hyperthyroidism, thyrotoxicosis) (Endocrine disorders) | 0 | 1 | 1
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 0 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0
Endocrine-Other (Specify) (Endocrine disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 1
Ocular/Visual-Other (Specify) (Eye disorders) | 1 | 0 | 0
Optic disc edema (Eye disorders) | 0 | 0 | 1
Retinal detachment (Eye disorders) | 3 | 1 | 1
Vision-flashing lights/floaters (Eye disorders) | 0 | 0 | 1
Distention/bloating, abdominal (Gastrointestinal disorders) | 0 | 1 | 0
Necrosis, GI - Ileum (Gastrointestinal disorders) | 0 | 1 | 0
Obstruction, GI - Small bowel NOS (Gastrointestinal disorders) | 1 | 0 | 0
Stricture/stenosis (including anastomotic), GI - Small bowel NOS (Gastrointestinal disorders) | 0 | 0 | 1
Ulcer, GI - Anus (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 2 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 2 | 1
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal-Other (Specify) (Gastrointestinal disorders) | 2 | 1 | 2
Heartburn/dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 1 | 1
Mucositis/stomatitis (functional/symptomatic) - Oral cavity (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 4 | 2
Pain - Abdomen NOS (Gastrointestinal disorders) | 3 | 3 | 4
Pain - Rectum (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 32 | 36 | 33
Death not associated with CTCAE term - Death NOS (General disorders) | 1 | 0 | 0
Death not associated with CTCAE term - Sudden death (General disorders) | 0 | 0 | 1
Edema: limb (General disorders) | 2 | 0 | 0
Flu-like syndrome (General disorders) | 0 | 1 | 0
Injection site reaction/extravasation changes (General disorders) | 0 | 0 | 1
Pain - Chest/thorax NOS (General disorders) | 2 | 1 | 2
Pain-Other (Specify) (General disorders) | 1 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 2 | 2
Hepatobiliary/Pancreas-Other (Specify) (Hepatobiliary disorders) | 3 | 2 | 4
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 1 | 5 | 1
Pain - Gallbladder (Hepatobiliary disorders) | 0 | 1 | 0
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 | 2 | 6
Allergy/Immunology-Other (Specify) (Immune system disorders) | 0 | 2 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils - Foreign body (e.g., graft, implant) (Infections and infestations) | 1 | 2 | 1
Infection (documented clinically or microbiologically) w/Grade 3 or 4 neutrophils -Skin (cellulitis) (Infections and infestations) | 0 | 1 | 0
Infection (documented clinically or microbiologically) w/Grade 3 or 4 neutrophils -Urinary tract NOS (Infections and infestations) | 1 | 0 | 0
Infection (documented clinically/microbiologically) w/Grade 3/4 neutrophils -Gallbladder (Infections and infestations) | 1 | 0 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils - Abdomen NOS (Infections and infestations) | 0 | 0 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Appendix (Infections and infestations) | 1 | 2 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Bladder (urinary) (Infections and infestations) | 1 | 1 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Kidney (Infections and infestations) | 0 | 1 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Lung (pneumonia) (Infections and infestations) | 2 | 3 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils - Pelvis NOS (Infections and infestations) | 0 | 0 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Skin (cellulitis) (Infections and infestations) | 4 | 10 | 12
Infection with normal ANC or Grade 1 or 2 neutrophils - Soft tissue NOS (Infections and infestations) | 0 | 1 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils - Urinary tract NOS (Infections and infestations) | 0 | 1 | 2
Infection with normal ANC or Grade 1 or 2 neutrophils - Vagina (Infections and infestations) | 1 | 0 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils - Wound (Infections and infestations) | 3 | 3 | 1
Infection with unknown ANC - Heart (endocarditis) (Infections and infestations) | 1 | 0 | 0
Infection with unknown ANC - Rectum (Infections and infestations) | 0 | 1 | 0
Infection with unknown ANC - Skin (cellulitis) (Infections and infestations) | 3 | 2 | 1
Infection with unknown ANC - Wound (Infections and infestations) | 0 | 0 | 1
Infection-Other (Specify) (Infections and infestations) | 0 | 1 | 2
Hemorrhage/bleeding associated with surgery, intra-operative or post-operative (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound complication, non-infectious (Injury, poisoning and procedural complications) | 0 | 1 | 1
Fracture (Injury, poisoning and procedural complications) | 8 | 8 | 12
Intra-operative injury - Vein NOS (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rash: dermatitis associated with radiation - Radiation (Injury, poisoning and procedural complications) | 2 | 0 | 1
Thrombosis/embolism (vascular access-related) (Injury, poisoning and procedural complications) | 17 | 17 | 7
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 1 | 3 | 2
AST, SGOT (serum glutamic oxaloacetic transaminase) (Investigations) | 1 | 1 | 0
Creatinine (Investigations) | 0 | 1 | 0
GGT (gamma-glutamyl transpeptidase) (Investigations) | 2 | 3 | 5
Leukocytes (total WBC) (Investigations) | 0 | 1 | 0
Weight loss (Investigations) | 0 | 2 | 2
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1 | 9 | 5
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 2 | 2 | 0
Iron overload (Metabolism and nutrition disorders) | 0 | 1 | 0
Pancreatic endocrine: glucose intolerance (Metabolism and nutrition disorders) | 3 | 14 | 3
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lumbar spine-range of motion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal/Soft Tissue-Other (Specify) (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3
Myositis (inflammation/damage of muscle) (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 3 | 2
Pain - Back (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain - Joint (Musculoskeletal and connective tissue disorders) | 64 | 55 | 119
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Hemorrhage, CNS (Nervous system disorders) | 0 | 1 | 0
CNS cerebrovascular ischemia (Nervous system disorders) | 4 | 1 | 3
Cognitive disturbance (Nervous system disorders) | 1 | 1 | 1
Dizziness (Nervous system disorders) | 3 | 0 | 5
Memory impairment (Nervous system disorders) | 0 | 0 | 1
Myelitis (Nervous system disorders) | 0 | 0 | 1
Neurology-Other (Specify) (Nervous system disorders) | 2 | 1 | 2
Neuropathy: cranial - CN V Motor-jaw muscles; Sensory-facial (Nervous system disorders) | 1 | 0 | 0
Neuropathy: cranial - CN VIII Hearing and balance (Nervous system disorders) | 0 | 1 | 1
Neuropathy: sensory (Nervous system disorders) | 1 | 5 | 4
Pain - Head/headache (Nervous system disorders) | 6 | 10 | 10
Pain - Neuralgia/peripheral nerve (Nervous system disorders) | 0 | 2 | 6
Syncope (fainting) (Nervous system disorders) | 1 | 2 | 4
Vasovagal episode (Nervous system disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 29 | 46 | 45
Mood alteration - anxiety (Psychiatric disorders) | 2 | 2 | 1
Mood alteration - depression (Psychiatric disorders) | 38 | 44 | 37
Psychosis (hallucinations/delusions) (Psychiatric disorders) | 0 | 0 | 1
Incontinence, urinary (Renal and urinary disorders) | 6 | 5 | 4
Obstruction, GU - Ureter (Renal and urinary disorders) | 0 | 1 | 4
Stricture/stenosis (including anastomotic), GU - Ureter (Renal and urinary disorders) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
Renal/Genitourinary-Other (Specify) (Renal and urinary disorders) | 49 | 19 | 11
Hemorrhage, GU - Ovary (Reproductive system and breast disorders) | 1 | 0 | 0
Hemorrhage, GU - Uterus (Reproductive system and breast disorders) | 5 | 1 | 3
Hemorrhage, GU - Vagina (Reproductive system and breast disorders) | 5 | 1 | 1
Stricture/stenosis (including anastomotic), GU - Uterus (Reproductive system and breast disorders) | 1 | 0 | 0
Irregular menses (change from baseline) (Reproductive system and breast disorders) | 4 | 2 | 0
Pain - Breast (Reproductive system and breast disorders) | 2 | 0 | 1
Pain - Ovulatory (Reproductive system and breast disorders) | 1 | 1 | 0
Pain - Pelvis (Reproductive system and breast disorders) | 1 | 0 | 0
Pain - Vagina (Reproductive system and breast disorders) | 14 | 22 | 19
Sexual/Reproductive Function-Other (Specify) (Reproductive system and breast disorders) | 0 | 2 | 2
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Obstruction/stenosis of airway - Bronchus (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pain - Pleura (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rash: erythema multiforme (e.g., Stevens-Johnson syndrome, toxic epidermal necrolysis) (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatology/Skin-Other (Specify) (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Pain - Skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus/itching (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Soft tissue necrosis - Thorax (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hematoma (Vascular disorders) | 1 | 0 | 0
Hot flashes/flushes (Vascular disorders) | 76 | 133 | 107
Hypertension (Vascular disorders) | 54 | 75 | 68
Thrombosis/thrombus/embolism (Vascular disorders) | 0 | 2 | 0
Vascular-Other (Specify) (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tamoxifen (N=1007) | T+OFS (N=1007) | E+OFS (N=1001)
Cardiac-ischemia/infarction (Cardiac disorders) | 1 | 2 | 5
Nausea (Gastrointestinal disorders) | 239 | 215 | 228
Fatigue (asthenia, lethargy, malaise) (General disorders) | 571 | 595 | 591
Injection site reaction/extravasation changes (General disorders) | 4 | 88 | 84
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 31 | 42 | 46
Fracture (Injury, poisoning and procedural complications) | 41 | 46 | 51
Thrombosis/embolism (vascular access-related) (Injury, poisoning and procedural complications) | 5 | 3 | 2
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 15 | 37 | 17
Pancreatic endocrine: glucose intolerance (Metabolism and nutrition disorders) | 15 | 21 | 28
Osteoporosis (Musculoskeletal and connective tissue disorders) | 123 | 198 | 316
Pain - Joint (Musculoskeletal and connective tissue disorders) | 631 | 700 | 778
Hemorrhage, CNS (Nervous system disorders) | 14 | 9 | 8
CNS cerebrovascular ischemia (Nervous system disorders) | 2 | 1 | 0
Insomnia (Psychiatric disorders) | 437 | 529 | 549
Libido (Psychiatric disorders) | 427 | 477 | 492
Mood alteration - depression (Psychiatric disorders) | 431 | 478 | 476
Incontinence, urinary (Renal and urinary disorders) | 156 | 180 | 120
Pain - Vagina (Reproductive system and breast disorders) | 224 | 240 | 290
Vaginal dryness (Reproductive system and breast disorders) | 421 | 500 | 541
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 486 | 621 | 566
Hot flashes/flushes (Vascular disorders) | 727 | 806 | 820
Hypertension (Vascular disorders) | 119 | 158 | 165

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2011-07-14): https://cdn.clinicaltrials.gov/large-docs/90/NCT00066690/Prot_001.pdf
  • Statistical Analysis Plan (2017-11-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT00066690/SAP_000.pdf